CLINICAL TRIAL: NCT00165724
Title: Alzheimer's Disease Long-term Follow-up Study (ALF Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKI-1002
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2010-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

INTERVENTIONS:
Drug: Donepezil Hydrochloride

SUMMARY:
Open study for efficacy and safety of donepezil treatment during 48 weeks

ELIGIBILITY:
Inclusion criteria

* Men or women aged 40 to 90
* Diagnosis of dementia according to DSM-IV
* Diagnosis of probable AD as defined by NINCDS-ADRDA criteria
* Mild to moderate AD at baseline, as defined by MMSE score of 10 to 26
* Patients were generally healthy and ambulatory or ambulatory aided
* Patients did not take acetylcholinesterase inhibitor 4 weeks before screening
* Patients have useful MRI results 3 months before screening

Exclusion

* If they have evidence of TIA or major infarction
* Epilepsy patients
* If they have evidence of other degenerative or psychiatric disorder, other serious disorder, alcoholism or drug abuse
* If they sensitive to acetylcholinesterase
* If they taken concomitant medication which were not allowed

Ages: 40 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2004-06-30 (Actual); Primary Completion 2006-07-31 (Actual); Study Completion 2006-12-31 (Actual)

PRIMARY OUTCOMES:
ADAS-cog

SECONDARY OUTCOMES:
MMSE, CDR, GDS, NPI, ADL, SSDQ

CONTACTS AND LOCATIONS:
Overall Officials: Jiheed Mun, Study Director — Eisai Korea Inc.
Locations (7):
- South Korea (7):
  - Bobath Memorial Hospital, Bundang
  - Bundang Seoul National University Hospital, Bundang
  - Changwon Fatima Hospital, Changwon
  - Yeungnam University Hospital, Daegu
  - Inha University Hospital, Incheon
  - Catholic University Hospital, Seoul
  - Eulji University Hospital, Seoul